CLINICAL TRIAL: NCT01937026
Title: A Study to Investigate the Potential Impact of Organic Anion Transporter 3 Inhibition by Probenecid on the Pharmacokinetics of Baricitinib (LY3009104) in Healthy Subjects
Brief Title: A Study of Baricitinib and Probenecid in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14604; I4V-MC-JAGG (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-09-03; First posted 2013-09-09 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — baricitinib; Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baricitinib (Experimental): Single oral dose of 4 milligrams (mg) baricitinib on Day 1
  Interventions: Drug: Baricitinib
- Baricitinib + Probenecid (Experimental): Oral doses of 1000 mg probenecid once daily on Days 3 through 7, with a single oral dose of 4 mg baricitinib co-administered on Day 5
  Interventions: Drug: Baricitinib; Drug: Probenecid

INTERVENTIONS:
Drug: Baricitinib — Administered orally
Drug: Probenecid — Administered orally
  Arms: Baricitinib + Probenecid

SUMMARY:
The purposes of this study are to assess how the body handles baricitinib when it is given with another drug called probenecid. The study doctor will measure the amount of baricitinib that is absorbed into the blood stream and the time that it takes to remove baricitinib from the body. The safety and tolerability of these drugs will be studied. The study will last about 18 days from the first dose to the end of the study (not including screening).

ELIGIBILITY:
Inclusion Criteria:

* Male participants: agree to use 2 reliable methods of birth control with female partners of childbearing potential during the study and for at least 3 months following the last dose of study drug
* Female participants: women not of childbearing potential due to surgical sterilization confirmed by medical history or menopause
* Have a body mass index of 18.0 to 29.0 kilograms per meter square (kg/m^2), inclusive
* Have clinical laboratory test results within the normal reference range
* Have normal renal function
* Have normal blood pressure and pulse rate

Exclusion Criteria:

* Are currently enrolled in a clinical trial or are concurrently enrolled in any other type of medical research
* Have completed or discontinued within the last 90 days from a clinical trial involving a study drug
* Are participants who have previously completed or withdrawn from this study or any other study investigating baricitinib, and have previously received baricitinib
* Have known allergies to baricitinib, probenecid, related compounds, or any components of the baricitinib or probenecid formulations, or history of significant atopy
* Have an abnormality in the 12-lead electrocardiogram (ECG)
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs;
* Have a history of or current gout or gouty arthritis
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Have a current or recent history of a clinically significant bacterial, fungal, parasitic, viral, or mycobacterial infection
* Have had symptomatic herpes zoster or herpes simplex infection within 90 days prior to the first dose
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C infection and/or positive hepatitis C antibody
* Show evidence of hepatitis B infection and/or positive hepatitis B surface antigen
* Are women who are lactating
* Intend to use over-the-counter or prescription medication (including salicylate drugs) and/or herbal supplements within 14 days prior to dosing and during the study or intended use of vitamin supplements from first dose of study drug until discharge from the Clinical Research Unit (CRU)
* Have consumed or intend to consume grapefruit or grapefruit-containing products within 7 days prior to the first dose and throughout the study
* Have used or intend to use any drugs or substances that are known to be substrates, inhibitors, or inducers of organic anion transporter (OAT)3 or cytochrome P450 (CYP) 3A4
* Have donated or lost blood of more than 500 milliliter (mL) within the last 3 months
* Have an average weekly alcohol intake that exceeds 28 units per week (males) and 21 units per week (females), or are unwilling to stop alcohol consumption from 48 hours prior to the first dose until discharge from the CRU at the end of study
* History of, in the opinion of the investigator, excessive methylxanthine use within the previous 6 months, such as greater than (>) 6 cups of coffee (or equivalent) per day
* Currently smoke more than 10 cigarettes per day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, 2-period, fixed-sequence study.
Groups:
- Baricitinib: 4 milligram (mg) baricitinib tablet administered orally, once, on Day 1 in Period 1 and on Day 5 in Period 2.
  1000 mg probenecid tablet administered orally, twice daily (BID), on Days 3 through 7 in Period 2.
Period: Period 1 (Day 1 Through Predose Day 3)
Arm/Group | Baricitinib
Started | 18
Received Baricitinib | 18
Completed | 18
Not Completed | 0
Period: Period 2 (At Dosing Day 3 Through Day 8)
Arm/Group | Baricitinib
Started | 18
Received Baricitinib | 18
Received Probenecid on Days 3 Through 7 | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Baricitinib: 4 mg baricitinib tablet administered orally, once, on Day 1 in Period 1 and on Day 5 in Period 2.
  1000 mg probenecid tablet administered orally, BID, on Days 3 through 7 in Period 2.
Arm/Group | Baricitinib
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 18

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Baricitinib
Time Frame: Days 1 and 5: predose of baricitinib, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 and 72 (Day 5 dosing only) hours postdose
Population: All enrolled participants who received study drug (baricitinib in Period 1 and baricitinib + probenecid in Period 2) and had PK data to calculate Cmax of baricitinib.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- Baricitinib: 4 mg baricitinib tablet administered orally, once, on Day 1 in Period 1.
- Baricitinib + Probenecid: 4 mg baricitinib tablet administered orally, once, on Day 5 in Period 2.
  1000 mg probenecid tablet administered orally, BID, on Days 3 through 7 in Period 2.
Arm/Group | Baricitinib | Baricitinib + Probenecid
Number analyzed (Participants) | 18 | 18
nanograms/milliliter (ng/mL) | 36.2 (22) | 37.3 (20)

2. Primary Outcome: PK: Area Under the Concentration Curve From Time 0 to Infinity [AUC (0-∞)] of Baricitinib
Time Frame: Days 1 and 5: predose of baricitinib, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 and 72 (Day 5 dosing only) hours postdose
Population: All enrolled participants who received study drug (baricitinib in Period 1 and baricitinib + probenecid in Period 2) and had PK data to calculate AUC (0-∞) of baricitinib.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | Baricitinib | Baricitinib + Probenecid
Number analyzed (Participants) | 18 | 18
nanograms*hour/milliliter (ng*h/mL) | 236 (22) | 480 (14)

ADVERSE EVENTS:
Time Frame: Baseline through study completion (up to Day 18).
Groups:
- Baricitinib: 4 mg baricitinib tablet administered orally, once, on Day 1 in Period 1.
  Adverse events are reported from baseline through predose on Day 3.
- Probenecid: 1000 mg probenecid tablet administered orally, BID, on Days 3 through 4 in Period 2.
  Adverse events are reported from postdose on Day 3 through predose on Day 5.
- Baricitinib + Probenecid: 4 mg baricitinib tablet administered orally, once, on Day 5 in Period 2.
  1000 mg probenecid tablet administered orally, BID, on Days 5 through 7 in Period 2.
  Adverse events are reported from postdose on Day 5 up to Day 18.
Arm/Group | Baricitinib | Probenecid | Baricitinib + Probenecid
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 3/18 | 3/18 | 8/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baricitinib (N=18) | Probenecid (N=18) | Baricitinib + Probenecid (N=18)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 6 (6)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days